CLINICAL TRIAL: NCT03525184
Title: Nutrition Intervention to Promote Immune Recovery From Sleep Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tracey Smith, Nutrition Scientist, United States Army Research Institute of Environmental Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-27HC
Record Dates: First submitted 2018-02-06; First posted 2018-05-15 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Sleep Restriction

STUDY DESIGN:
Intervention Model Description: Participants will undergo the study during normal sleep, sleep restriction without the multi-nutrient beverage and sleep restriction with the multi-nutrient beverage
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal sleep (Placebo Comparator): A normal sleep condition and the placebo treatment (0.9 g protein/kg body weight/day + placebo beverage; NS)
  Interventions: Other: Placebo beverage
- 72-h Sleep restriction with placebo beverage (Placebo Comparator): Sleep restriction (72-h with 2-h of sleep per night) and the placebo treatment (0.9 g protein/kg body weight/day + placebo beverage; SR),
  Interventions: Other: Placebo beverage
- 72-h Sleep restriction with multi-nutrient beverage (Experimental): Sleep restriction (72-h with 2-h of sleep per night) and the experimental treatment (1.5 g protein/kg body weight/day + multi-nutrient beverage; SR+).
  Interventions: Other: Additional protein and multi-nutrient beverage

INTERVENTIONS:
Other: Additional protein and multi-nutrient beverage — During SR+, participants will consume a multi-nutrient beverage and additional protein (~1.5 grams·kg-1 body weight·day-1 versus the lower end of MDRI of ~0.9 grams·kg-1 body weight·day-1) during and after the period of sleep restriction. The multi-nutrient beverage contains arginine, glutamine, vits C & D, zinc and omega-3 fatty acids (DHA and EPA).
  Arms: 72-h Sleep restriction with multi-nutrient beverage
Other: Placebo beverage — The placebo beverage (NS and SR) will be composed of a commercially-available artificially sweetened (e.g., containing aspartame, splenda or another artificial sweetener) beverage powder base and grapefruit extract (i.e., naringen) and/or quinine (i.e., a common ingredient found in tonic water).
  Arms: 72-h Sleep restriction with placebo beverage; Normal sleep

SUMMARY:
Physical and psychological stress on Warfighters during training and operational missions can suppress immune responsiveness. Skin wound models can be used to detect changes in immune function. Investigators have recently demonstrated that relatively modest sleep disruption degrades immune response at the site of the disrupted skin barrier and delays the initial restoration of the skin barrier. Provision of additional protein and a multi-nutrient beverage during and after sleep restriction seems to mitigate decrements in local immune function, without producing detectable effects on initial restoration of the skin barrier. However, the prior work used a parallel-group study design and inter-subject variability may have made it more difficult to detect significant differences in skin barrier restoration between participants receiving the nutrition intervention versus those receiving the placebo. Therefore, the purpose of the proposed cross-over study is to test the efficacy of a multi-nutrient beverage and additional protein (1.5 g protein per kg body weight versus 0.9 g protein per kg body weight) on immune function and the initial restoration of the skin barrier consequent to an operational stressor (i.e., 72-h sleep restriction). The effect of sleep restriction on a friend-foe marksmanship task, flow state, and measures of cognitive and neuromotor performance, will be investigated as a sub-study (Appendix A). Additionally, the effects of sleep restriction on appetite physiology, eating behaviors and intestinal permeability will be tested. Research will be conducted in a laboratory environment using male and female Soldiers from the human research participant detachment (NSRDEC), or Soldiers or civilians at NSRDEC and/or USARIEM. Participants in the study described herein (n = 20) will be exposed, in a single-blind, cross-over design to a ~72 hour normal sleep control phase, and to 2 periods of ~72 hours of sleep restriction (monitored in laboratory with ~2-h sleep per night) during which time eight blisters will be induced via suction on participant's forearm and the top layer of blisters will be removed to reveal the dermal layer of skin. In the normal sleep trial, participants will consume ~0.9 g protein per kg body weight per day and a placebo beverage during (3 days). In the first sleep restriction trial, participants will consume ~0.9 g protein per kg body weight per day and a placebo beverage during (3 days) and after (5 days) sleep restriction; and, in the second sleep restriction trial (after at least two weeks wash-out) participants will instead consume ~1.5 g protein per kg body weight and a multi-nutrient beverage (arginine: 20 g·d-1, glutamine: 30 g·d-1, zinc sulfate: 24 mg·d-1, vitamin C: 400 mg·d-1, vitamin D3: 800 IU·d-1 and omega-3 fatty acids: 1 g·d-1). Outcome measures include immune function (e.g., circulating markers of inflammation, cytokines at the blister site, and secretory immunoglobin A), skin barrier restoration time (by transepidermal water loss), subjective appetite ratings, appetite-mediating hormone concentrations, food preferences and cravings, gut microbiota composition, and intestinal permeability. Findings from this study will determine if a nutritional intervention attenuates the loss of immune responsiveness to a military relevant stressor (i.e., sleep restriction), and will determine the effects of acute sleep restriction on appetite, gut microbiota composition, and intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

Active duty military personnel and civilians with prior rifle marksmanship experience, and who sleep between 7 and 9 hours per night at least 5 days per week, and are between the ages of 18 and 45 will be invited to participate in this study.

Exclusion Criteria:

Potential participants will be excluded from participation if they:

* are under the age of 18 or over the age of 45;
* have a tattoo on either forearm; are taking nonsteroidal anti-inflammatory drugs (e.g., Advil), aspirin, lipid-lowering drugs or corticosteroids; pregnant or lactating; are immune-compromised (e.g., chemotherapy or radiation treatment);
* are suffering from an autoimmune disease (e.g., lupus);
* recovering from a surgery within the past 6 months; have an injury that will prevent physical activity;
* have a recent eye injury (within the past 6 months) or have had eye surgery within the past year, have doctor-diagnosed dry eye syndrome;
* have a history of cardiovascular or metabolic disease; are suffering from sleep apnea; have a history of psychiatric disorder requiring hospitalization or have taken psychiatric medication (e.g., anti-depressants or anti-anxiety medication) within the past three years for any length of time;
* are suffering from any neurological disorder (e.g., epilepsy or other seizure disorder, narcolepsy or other sleep disorders, or multiple sclerosis);
* have a history of gastrointestinal disease (such as celiac disease, irritable bowel syndrome, colitis, and Crohn's disease), have taken oral antibiotics within the 3 months prior to study participation;
* and have a Body Mass Index (BMI) ≥ 30;
* have speech, facial or muscle disorder or injuries preventing them from producing a normal range of hand or finger motion.
* Participants will be asked not to sign the consent form if they regularly (more than 2 days per week) sleep less than 7 hours or more than 9 hours per night; or, take a nap 3 or more days per week.
* Potential participants will also be excluded from participation if they will feel uncomfortable handling a weapon, shooting at silhouette targets, have an injury that will impair firing a rifle, have ever been diagnosed with post-traumatic stress disorder, are unable to distinguish the color "red" from the color "black", or have a bowel movement less frequently than every-other-day.
* Potential participants also must agree to abstain from smoking, chewing or vaping tobacco or nicotine-containing products during the live-in portions of the study.
* Participants must be able to speak and read English fluently and will require a general medical clearance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Partial skin barrier restoration | up to 10 days
  Partial restoration of the skin barrier (i.e., to demonstrate initial phases of the wound healing process)

SECONDARY OUTCOMES:
Cytokine response of local wound fluid (e.g., IL-6, IL-8, TNF-a) | 4, 7, 24, 48, 72 and 96-hours
  Immune response of blister fluid

OTHER OUTCOMES:
Lactulose:mannitol ratio of urine | 5-h
  Determining the effects of acute sleep restriction and multi-nutrient supplementation on intestinal permeability using dual sugar test (i.e., lactulose and mannitol).
Appetite ratings | Throughout study participation (~68 days)
  Appetite ratings are calculated from participants using a visual analogue scale, wherein the participant places a slash mark across a line spanning 100 cm (with one end being extremely hungry and the other end being extremely full).
Energy consumption | Throughout study participation (~68 days)
  Energy consumption during ad libitum meals
Eating rate | Throughout study participation (~68 days)
  Eating behavior determined by measuring eating rate using Madometer device during multiple meals over the course of the 68-day study
Marksmanship accuracy | 0, 24, 48 and 72-hours
  Accuracy of discriminating friend and foe, using simulated marksmanship to determine effects of sleep restriction marksmanship performance
Marksmanship speed | 0, 24, 48 and 72-hours
  Speed of trigger pull using simulated marksmanship to determine effects of sleep restriction marksmanship performance

CONTACTS AND LOCATIONS:
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith TJ, Wilson M, Whitney C, Fagnant H, Neumeier WH, Smith C, Heaton KJ, Cho E, Spielmann G, Walsh NP, Karl JP. Supplemental Protein and a Multinutrient Beverage Speed Wound Healing after Acute Sleep Restriction in Healthy Adults. J Nutr. 2022 Jun 9;152(6):1560-1573. doi: 10.1093/jn/nxac064. PMID 35285906
- [Derived] Radcliffe PN, Whitney CC, Fagnant HS, Wilson MA, Finlayson G, Smith TJ, Karl JP. Severe sleep restriction suppresses appetite independent of effects on appetite regulating hormones in healthy young men without obesity. Physiol Behav. 2021 Aug 1;237:113438. doi: 10.1016/j.physbeh.2021.113438. Epub 2021 Apr 30. PMID 33940082